CLINICAL TRIAL: NCT01655537
Title: Cognitive Dysfunction in Fibromyalgia Patients: Specific Neuro-psychological Dysfunctions, Psychiatric Comorbidity and Integrative Assessments
Brief Title: Cognitive Dysfunction in Fibromyalgia Patients
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Rena Cooper, Psychiatric Outpatient Clinic-Head, Hadassah Medical Organization
Other Study IDs: COG-FM-HMO-CTIL
Record Dates: First submitted 2012-07-31; First posted 2012-08-02 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; cognitive dysfunction
MeSH Terms: conditions — Fibromyalgia; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Fibromyalgia is a common rheumatologic disorder. Many patients complain of cognitive dysfunction as part of their symptoms.

The investigators aim to assess this cognitive dysfunction through extensive neuro-cognitive testing.

DETAILED DESCRIPTION:
Cognitive dysfunction in Fibromyalgia patients: specific neuro-psychological dysfunctions, psychiatric comorbidity and integrative assessments - Can the investigators help them?

Scientific and Technological Background

1. General Clinical characteristics FM is a common rheumatologic disorder (ranges from 2%-12% in the general population) with complex symptom presentation that include: chronically painful, soft tissue pain. Those affected suffer widespread pain and tenderness at anatomically defined tender points in soft tissue musculoskeletal structures. Associated symptoms include depression, anxiety, fatigue, sleep disturbances, and other somatic complaints (headaches, irritable bowel or bladder, morning stiffness, dysesthesia) and severe cognitive impairment. Cognitive impairment in FM has both subjective elements: "forgetfulness", "concentration difficulties" or "a failing memory".
2. Cognitive impairment in FM 2.1 Subjective Cognitive impairment in FM The subjective cognitive impairments have been described in several studies. Zachrisson and colleagues reported a 95% incidence rate for ''Concentration Difficulties'' and a 93% incidence rate for ''Failing Memory'' on their Fibro-Fatigue scale. Additionally, patients who have FM report more cognitive problems and dissociative states than other rheumatology patients. Arnold and colleagues reported the results of patient focus groups that assessed important symptoms and the impact of these symptoms from a patient perspective. Patients reported that memory and concentration problems were very disruptive-affecting their ability to express themselves due to word-finding difficulties, their ability to organize and plan ahead, their ability to respond quickly to questions, and their ability to drive.

   2.2 Objective Cognitive impairment in FM Objective cognitive dysfunction is assessed through a broad range of neuro-cognitive testing. The mechanisms found to have the most marked impairment in FM are: working memory, followed by episodic memory and access to semantic memory. In addition findings points to a particular difficulty in dealing with distracting information so that patients have an enhanced sensitivity to distraction and difficulty in filtering sensory stimuli.

   2.2.1 Working memory Working memory is a system of short-term memory storage system (on the order of seconds) combined with other mental processes, that allows for example, to briefly remember two numbers and add them together mentally. A quick assessment of working memory function is: how many digits an individual can listen to and then repeat in backward order. Working memory is a basic cognitive mechanism that underlies successful performance on many other cognitive tasks. There are now several studies that have reported impairment in this important cognitive function in subjects who have FM, using a variety of different tests of working memory.

   (A) Paced auditory serial attention test (PASAT): Most studies using the PASAT found lower performance in subjects who have FM compared with controls although Suhr did not find differences.

   (B) Auditory Consonant Trigram (ACT) test: Both Leavitt and Katz and Dick and colleagues found that subjects who have FM recalled fewer of the trigrams correctly, and many performed in the impaired range compared with the control participants.

   (C) Reading Span Task is a working memory test used extensively to study age-related decline in working memory : Park and colleagues and Dick and colleagues found that subjects who have FM perform more poorly than age-matched controls. Furthermore, Park and colleagues found that performance in the subjects who have FM was not different from control subjects who were 20 years older.

   (D) Test of Everyday Attention (TEA) showed that subjects who have FM had lower scores on the working memory component of the TEA.

   The wide variety of working memory tests that demonstrate lower performance in FM is striking, suggesting that this impairment is quite robust. Because deficits in working memory ability have repercussive effects on other aspects of cognition, a small deficit in working memory may have a large impact on performance on complex tasks. A busy work environment requires an employee to hold some information in mind while using that information for further processing.

   2.2.2 Episodic Memory

   Episodic memory refers specifically to the ability to remember specific events or episodes from one's life (Remembering your first day at school or the name of your teacher). Several researchers have found deficits in episodic memory in subjects who have FM using a wide variety of standardized neuro-psychological tests and some laboratory tests. Several of these results are presented:

   (A) Grace and colleagues found significant differences on the general memory, verbal memory, and delayed recall components of the Wechsler Memory Scale-Revised (WMS-R), but not on the visual memory or attention/concentration components.

   (B) Leavitt and Katz found that subjects who have FM, performed slightly below the norm on logical memory and paired associates.

   (C) Glass and colleagues found that subjects who have FM recalled fewer words in a list learning task, and their memory was most impaired when combined with a distracting secondary task at both list learning and recall.

   These and other findings suggest a mild impairment in episodic memory in FM patients. However, the results of episodic memory testing do not seem to be as robust as the working memory results. In addition, Leavitt and Katz suggest that memory function in FM may be strong enough to perform well under ideal conditions (neuro-cognitive testing), but performance decrements may be observed in the presence of distraction.

   2.2.3 Semantic memory Semantic memory is the knowledge of words and facts that have been learned, such as knowing that eggs and milk are sources of protein (21). It can be measured in a number of ways. One method uses verbal fluency to measure how quickly and efficiently stored knowledge about words can be accessed. Several studies indicate impairment in verbal fluency in FM.

   (A) Park and colleagues found that FM subjects produced fewer words during a fluency test compared to age-matched controls.

   (B) Landro and colleagues and Munguia-Izquierdo and Legaz-Arrese) also reported similar findings.

   (C) Suhr did not find any difference between subjects who have FM and controls on a fluency test.

   (D) Park and colleagues and Glass and colleagues also found that FM subjects perform more poorly than education- matched controls on tests of vocabulary (another test of semantic memory).

   (E) Leavitt and Katz reported a naming speed deficit in FM, consistent with the verbal fluency results.

   Thus, patients who have FM seem to have a deficit in accessing stored knowledge. This deficit can make it difficult for patients to think quickly and to come up with the right word for a given situation. Several patients indicated this kind of word-finding difficulty while interviewed in a patient focus group.

   2.2.4 Attention, concentration and executive functions Attention and working memory are very closely linked because attention mechanisms are used to control the items that are accessed, stored and processed in working memory. The working memory problems found in FM patients may be due to the management of the contents of working memory, using attention and concentration.

   (A) Leavitt and Katz suggest that the cognitive impairment in FM patients is more prominent on tasks where distraction from a competing source of information was prominent (PASAT, ACT) in contrast to tasks without distraction (digit span, logical memory, paired associate).

   (B) Others found that distraction reduced memory abilities in FM subjects when attention was divided during the learning.

   (C) Dick and colleagues reported that FM subjects perform at a lower level than healthy controls on the TEA test of attention.

   (D) In a recent study performed by Verdejo-Garcia and colleagues, executive functions and decision making were assessed in FM using the Wisconsin Card Sorting Task (WCST) and the Iowa Gambling Task (IGT). FM subjects achieved a lower number of categories and made more non-perseverative errors on the WCST. On the IGT, subjects who have FM showed an altered learning curve that suggested a hypersensitivity to reward. These new data on executive functions fit well with the attention control difficulties.

   Dealing with distraction or controlling what is attended to, are particular problems in FM and come under the category of executive functions. Planning a goal-directed behavior and monitoring it are also under that category. Taken together, these results strongly suggest that executive functions are impaired in FM patients.
3. Possible causes of cognitive dysfunction in FM

   3.1 Other mental symptoms Mental symptoms such as depression and anxiety are suspected to play an important role in the development of cognitive dysfunction in FM. Sephton et al found depressive symptoms to be negatively correlated with verbal recall and Surh found them to be related to memory. Grace et al reported an association between anxiety and measures of memory and concentration. An important question was whether these dysfunctions remained after correcting for depression and anxiety. Indeed, Dick et al reported a significant difference between controls and FM patients even after correcting for depression and anxiety. Park et al and Verdejo-Garcia et al did not find a significant correlation between these mental symptoms and performance on cognitive measures. In summary, depressive symptoms and anxiety can contribute to cognitive dysfunction but they do not entirely explain it.

   3.2 Fatigue and sleep disturbances Impaired sleep is known to negatively affect cognitive performance. Cote -Moldofsky and Suhr attempted to explain the possible relationship between altered sleep architecture and cognitive performance. Suhr specifically reported that fatigue was related to psychomotor speed. Dick et al reported that the differences between control and FM patients remained even after controlling for sleep disturbances. Thus, as is the case in mental symptoms, fatigue and sleep disturbances can not fully explain the cognitive deficit in FM patients.

   3.3 Pain Chronic pain is known to negatively affect cognitive performance. Various cognitive tasks including, impaired attention, impaired learning on a decision-making task and an attentional bias to pain-related stimuli, were found in chronic pain patient and in FM patients specifically. These patients were found to selectively attend to pain words. In many studies of FM patients specifically, self-reported levels of pain were associated with cognitive performance. These suggest that pain in itself may disrupt the normal function of attention. As apposed to the case with depression, anxiety and sleep disturbances, Dick et al, observed that the differences between controls and FM patients cognitive functions disappeared when controlled for pain.
4. Recent experience in our psychiatric clinic Over the past few months the investigators have been evaluating FM patients for cognitive dysfunction. Nearly 10 patients have undergone the above mentioned extensive assessment. In our assessment the investigators also added a more specific assessment of executive function; the "six elements" task. This task directs participants to perform several tasks while under both a time limitation and under specific rules. Thus, they are required to use: planning and organization, initiation, and monitoring. These processes are usually not taken under consideration during formal neuro-psychological tests because of their very structured nature. Our preliminary findings suggest that fibromyalgia patients show a pattern of executive dysfunction compared to the healthy population. The investigators hypothesize a similar pattern will be found in our more extensive research and suggest that significant executive dysfunction lie in the basis of cognitive dysfunction found in fibromyalgia patients.
5. Cognitive rehabilitation - Treatment options Cognitive rehabilitation, a behavioral treatment approach for individuals with cognitive dysfunction, is designed to reduce functional impairment and increase engagement in daily adaptive activities; vocational, social, and adaptive daily living skills. Originally developed to improve cognitive functioning after traumatic brain injury (TBI), cognitive rehabilitation programs have recently been adapted for other neurological conditions. Subsets of cognitive training programs have been developed to target improvement in specific cognitive domains including: attention, working memory, and executive functioning, which are all essential cognitive skills to complete daily living tasks.

For example, TBI patients' who underwent attention training, consisting of direct attention and metacognitive training to promote development of compensatory and problem solving strategies, showed improvement on complex attention measures. When it comes to mild memory impairment, compensatory strategies are recommended. Adults with chronic TBI, who were trained to use compensatory strategies for personally-relevant memory problems through errorless learning or didactic strategy instruction, reported greater use of strategies after training.

Metacognitive training (self monitoring and self regulation) for executive functions include problem solving strategies with application to everyday activities. The awareness training protocol incorporates feedback to increase participants' awareness of their abilities, with experiential exercises requiring participants to predict, self-monitor, and self-evaluate their performance. Improvement in awareness, performance of everyday tasks and overall function were evident for both TBI and stroke patients.

Cognitive decline and executive dysfunction are also common among Parkinson's disease patients. As in FM, executive dysfunction/attention and memory impairment are the most prevalent deficits reported. A computerized cognitive rehabilitation program focused on improving attention, abstract reasoning, and visuospatial abilities showed PD patients had significantly improved verbal fluency, immediate and delayed logical memory, and visuospatial reasoning compared with their baseline assessments; these gains were maintained after 6 months. Improvement on measures of executive skills were shown after completing an intervention consisted of in-person training with practice exercises and worksheets on attention tasks. Daily at-home practice exercises were also encouraged.

Similar cognitive impairment is also common among multiple sclerosis (MS) patients, reporting mainly attention and memory complaints. In a double-blinded, randomized, placebo controlled trial of an intervention to improve learning and memory, MS patients were taught to use a modified "story memory technique" which used context and imagery to improve learning and, therefore, recall. Participants who had moderate to severe learning impairments showed a significant improvement in learning abilities. The use of the modified story memory technique is recommended as a practice guideline for the remediation of learning and memory in MS patients.

In summary:

Altogether, these reports demonstrate quite conclusively the salience of cognitive dysfunction and its impact on daily life for patients who have FM. Comorbid symptoms (depression, anxiety, fatigue and disturbed sleep) can negatively impact on cognitive function, but can not fully explain the findings. In one study, pain did have a robust effect on cognitive function and could explain the dysfunction found in FM. There is a need to further assess cognitive function in FM along with the possible comorbid symptoms. Based on our preliminary findings there is also a need to broaden assessment of executive functions. In addition, cognitive rehabilitation has proved to be successful in a variety of conditions involve cognitive impairment. One may suggest that if a specific cognitive impairment pattern can be identified in FM patients, a cognitive rehabilitation plan can then be tailored to fit these patients' needs.

Research Objectives

The objects of the proposed research are to perform:

1. A broad neuro-cognitive testing battery on a large population of Fibromyalgia patients. Previous testing did not fully evaluate executive functions; therefore the investigators are adding specific testing for these functions.
2. A broad assessment for Axis I psychiatric co-morbidity in the FM population.
3. A broad assessment for FM additional symptoms: depressive symptoms, anxiety, fatigue, pain, sleep disturbances.
4. An attempt to identify "pure" cognitive deficits that are unique to FM patients and can be directly attributed to FM. Therefore, possible correlation between neuro-cognitive impairments, Axis I psychiatric diagnoses, additional FM symptoms and motivation levels will be performed and data will be analyzed while controlling for these confounders.
5. Develop a cognitive rehabilitation program based on the cognitive dysfunction the investigators discover in the study.
6. Based on the cognitive dysfunction the investigators discover in the study the investigators hope to compile a shorter neuro-cognitive battery for clinical use in FM patients.

   * Research Plan________________________________ A. Methodology and plan of operation

A.1 Overview This is an open study in which a large number of fibromyalgia patients will undergo an extensive neuro-cognitive assessment. All consenting participants will be assessed using well validated neuro-cognitive tests. Current Axis I, psychiatric comorbidity will be assessed using a well validated questionnaires. Finally, other symptoms associated with FM will also be assessed (depression, anxiety, fatigue, sleep and pain) with the appropriate rating scales. This assessment will be performed by a trained neuro-psychologist and will take place in the psychiatric clinic during two consecutive sessions.

A.2 Patient selection A.2.1 Inclusion criteria 1. Primary fibromyalgia as defined by the American College of Rheumatology 2. Age 18-70 years 3. Male or female 4. Competent and willing to give written informed consent 4.A.2.2 Exclusion Criteria

1. History of head trauma
2. Any significant neurological disorder that may confound neuro-cognitive testing

A.3 Sample size The investigators plan to recruit 100 fibromyalgia patients over a period of 18 months. This is an exceptionally large number of patients. It is large enough to fully assess the neuro-cognitive dysfunction in FM patients while controlling for psychiatric symptoms and other additional FM symptoms.

A.4 Assessment of patients

A.4.1 Neuro-cognitive testing

1. Adult Intelligence Scale - WAIS III - relevant subtests from Wechsler Adult Intelligence Scale-III 2. Verbal memory - Rey AVLT - adapted for Hebrew speakers 3. Motor ability and visual memory

1. Rey Complex Figure Test
2. Bender Gestalt II 4. Executive function assessment

<!-- -->

1. Wisconsin Card Sorting Test
2. Verbal Fluency - adapted for Hebrew speakers
3. Six Elements
4. Clock drawing test

   A.4.2 Psychiatric rating scales and questionnaire

   Axis I comorbidity -general -

   1. Structured Clinical Interview for Axis I DSM-IV disorders (SCID) - Hebrew version Depression
   1. Hamilton Depression Scale, 21 items (HAM-D)
   2. Beck Depression Inventory (BDI)
   3. 100mm Visual Analog Scale (VAS) for depression Anxiety

   1. Hamilton Anxiety Scale (HAM-A)

   A.4.3 Assessment of associated symptoms; FM, Pain, fatigue and sleep disturbances

   Fibromyalgia severity
   1. Fibromyalgia Impact Questionnaire (FIQ)-Hebrew version
   2. Fibromyalgia rating scale (FRS)
   3. Clinical Global Impression of Severity (CGI) (for fibromyalgia) Pain

   <!-- -->

   1. 100mm Visual Analog Scale (VAS) for pain
   2. Brief Pain Inventory (BPI) Fatigue

   1. Fatigue Severity Scale 2. Brief Fatigue Inventory Sleep disturbance

   1. Insomnia Severity Scale

   B. Time schedule The investigators plan on recruiting the patients over a period of 18 months. The analysis of the data will take a further 6 months.

   C. Expected results The investigators expect to find extensive but specific pattern of cognitive dysfunction in the FM patients, compared to the norms found in the healthy population. The investigators expect to find cognitive dysfunction in the field of: working memory, episodic memory, semantic memory. The investigators are expanding the assessment to include executive functions and expect to find significant dysfunction in this area. The investigators do expect to find psychological factors such as depression and anxiety and additional FM symptoms such as pain and fatigue. The investigators mean to control for these symptoms in order to expose the "pure" cognitive dysfunction characteristic of FM, that which can not be explained by these active symptoms.

   D. Significance FM is a common disabling disorder with many complex symptoms. Evidence continues to mount that cognitive dysfunction is a real and troubling symptom with working memory, episodic memory and semantic memory mostly affected. In addition, FM patients seem particularly sensitive to distraction and in our preliminary data they appear specifically to have executive dysfunction. This study aims to broadly assess neuro-cognitive function in FM patients for possible neuro-cognitive deficits with a specific focus on executive functions.

   Since Axis I psychiatric disorders, mental symptoms (depression and anxiety) and additional FM symptoms (fatigue, pain and sleep disturbances) may all affect cognitive function, the investigators will also assess these factors. In the analysis of our expected data the investigators will "control" for these possible confounders in hope of finding a unique neuro-cognitive dysfunction pattern specific for FM patients. The investigators than intend on compiling a shorter, "user friendly", neuro-cognitive battery, that may serve clinicians in their routine assessment of FM patients.

   The investigators aim to develop a cognitive rehabilitation program that will specifically address the cognitive dysfunction the investigators expect to discover in this study. Munguia-Izquierdo and Lagaz-Arrese found that aquatic therapy (exercise in warm water) indirectly improved many symptoms in FM, including cognitive function. Leavitt and Katz found that rehearsal helped subjects with FM overcome the effects of distraction in a memory test. Based on these studies, but more on the extensive knowledge from cognitive rehabilitation programs in other clinical states, the investigators are determined to develop our own cognitive rehabilitation program that will supplement other pharmacological and non-pharmacological interventions in FM patients. By this the investigators will offer a unique and novel intervention for Fm patients.

ELIGIBILITY:
Inclusion Criteria:

1. Primary fibromyalgia as defined by the American College of Rheumatology
2. Age 18-70 years
3. Male or female
4. Competent and willing to give written informed consent

Exclusion Criteria:

1. History of head trauma
2. Any significant neurological disorder that may confound neuro-cognitive testing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: fibromyalgia patients
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2012-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: RENA COOPER-KAZAZ, Dr., Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization-PSYCHIATRIC CLINIC, Jerusalem, Israel